CLINICAL TRIAL: NCT06207474
Title: A Study on BReast Cancer Patient Care Using chAtbot and Video Education for Radiation Therapy (BRAVE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 4-2022-0044
Record Dates: First submitted 2023-12-08; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Videotape Recording; Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video + Chatbot (Other)
  Interventions: Other: Video + Chatbot
- Video + Paper (Other)
  Interventions: Other: Video + Paper
- Paper + Chatbot (Other)
  Interventions: Other: Paper + Chatbot
- Paper + Paper (Other)
  Interventions: Other: Paper + Paper

INTERVENTIONS:
Other: Video + Chatbot — Participants will receive detailed information about the radiation therapy process, potential side effects, frequently asked questions, and aftercare instructions using a combination of educational videos and interactive chatbot sessions.
  Arms: Video + Chatbot
Other: Video + Paper — Participants will receive detailed information about the radiation therapy process, potential side effects, frequently asked questions, and aftercare instructions using a combination of educational videos and paper materials.
  Arms: Video + Paper
Other: Paper + Chatbot — Participants will receive detailed information about the radiation therapy process, potential side effects, frequently asked questions, and aftercare instructions using a combination of paper materials and interactive chatbot sessions.
  Arms: Paper + Chatbot
Other: Paper + Paper — Participants will receive detailed information about the radiation therapy process, potential side effects, frequently asked questions, and aftercare instructions using paper materials.
  Arms: Paper + Paper

SUMMARY:
This randomized trial explored whether digital media (videos and chatbots) used for patient education could more effectively reduce anxiety in breast cancer patients during radiation therapy, compared to traditional paper-based methods. Post-surgery breast cancer patients scheduled for radiation therapy were assigned to groups receiving treatment information through different media combinations. The study aimed to assess whether these modern tools more effectively ease anxiety, thus potentially improving patient compliance and treatment experience.

DETAILED DESCRIPTION:
This study evaluates the impact of patient management and information provision using educational videos and chatbots on patient experience, satisfaction, and patient psychology in the breast cancer radiation treatment process.

The experiment is designed as (2 (with or without using chatbot) X 2 (with or without using video) to distinguish groups.

There is no separate treatment intervention in addition to use chatbot and video utilization.

ELIGIBILITY:
Inclusion Criteria:

1. A breast cancer patient scheduled for radiation therapy after radical surgery.
2. Subjects must have the cognitive ability to use smartphone.
3. Age ≥ 20 year old

Exclusion Criteria:

1. Patients with visual or auditory impairment.
2. Subjects do not consent to participate in this study.
3. Pregnancy, fetus, newborn, underage
4. Age ≥ 75 year old

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
APAIS(Amsterdam Preoperative Anxiety and Information Scale) | baseline, before radiation therapy, after all radiation, an average of 1 month
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS): The APAIS consists of six self-reported items, primarily assessing anxiety associated with anesthesia and surgery.

SECONDARY OUTCOMES:
STAI-X(State-Trait Anxiety Inventory for Adults) | baseline, before radiation therapy, after all radiation, an average of 1 month
  The STAI is a widely recognized self-report instrument for gauging anxiety levels.
LASA(Linear Analog Scale Assessments) | baseline, before radiation therapy, after all radiation, an average of 1 month
  LASA is a tool to measure a patient's self-assessment of various aspects of their health and wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Bae Kim, Principal Investigator — Yonsei Cancer Center
Locations (1):
- Yonsei Cancer Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No